CLINICAL TRIAL: NCT04828174
Title: The Safety and Clinical Efficacy of Human TRBC1 CAR-T Cell Therapy for Patients With Relapsed/Refractory TRBC1 Positive T Cell Hematological Maliganacies
Brief Title: Anti-TRBC1 CAR-T Cell Therapy in Patients With TRBC1 Positive T Cell Malignancies
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: The trial was suspended due to the inability to enroll qualified participants
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Xianmin Song, MD, principal investigator, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHYSXY-202101-CART
Record Dates: First submitted 2021-03-31; First posted 2021-04-01 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Peripheral T Cell Lymphoma; Angioimmunoblastic T-cell Lymphoma; Anaplastic Lymphoma; Acute T Cell Leukemia; T-lymphoblastic Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral; Immunoblastic Lymphadenopathy; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- anti-TRBC1 CAR-T cell (Experimental): Administration with anti-TRBC1 CAR-T cells in the relapsed/refractory T cell hematological malignancy patients.
  Interventions: Drug: anti-TRBC1 CAR-T cell therapy

INTERVENTIONS:
Drug: anti-TRBC1 CAR-T cell therapy — TRBC1 positve patients with relapsed or refractory T cell malignacy will receive CAR-T cell therapy targetting TRBC1

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of CAR T cell treatment targeting TRBC1 in patients with relapsed or refractory TRBC1 positive T-cell hematological maliganacies

ELIGIBILITY:
Inclusion Criteria:

(1)18 to 70 Years Old, Male and female; (2) Expected survival > 12 weeks; (3) ECOG score 0-2; (4) Confirmed diagnosis of acute T cell leukemia and screened for TRBC1 positive, including following conditions:

1. Patients who do not get a CR with ≥2 prior lines of therapy
2. Those who achieves CR, but have a early relapse(<12months),or a late relapse (>=12months) failing to acheive a CR after 1 line salvage chemotherapy
3. For any Patiens failed ASCT/allo-SCT (5) Relapsed and refractory patients with diagnosis of T cell lymphoma have had≥2 prior lines of therapy,including:

a. Peripheral T cell lymphoma NOS, or b. Angioimmunoblastic T cell lymphoma, or c. Anaplastic large cell lymphoma (6) Confirmed T lymphoblatic lymphoma

1. Patients who do not get a CR with ≥2 prior lines of therapy
2. Relapsed patients failing to acheive a CR after 1 line salvage chemotherapy
3. For any Patiens failed ASCT/allo-SCT (7) The venous access required for collection can be established and mononuclear cell collection can be determined by the investigators; (8) Liver, kidney and cardiopulmonary functions meet the following requirements:

a. Ccr≥60mL/min(Cockcroft Gault) b. Left ventricular ejection fraction >50%; c. Baseline oxygen saturation>92%; d. Total bilirubin ≤ 1.5×ULN; e. ALT and AST ≤ 3×ULN; (9) Able to understand and sign the In

Exclusion Criteria:

1. Malignant tumors other than acute lymphoblastic leukemia within 5 years prior to screening, in addition to adequately treated cervical carcinoma in situ, basal cell or squamous cell skin cancer, localized prostate cancer after radical resection, and ductal carcinoma in situ after radical resection;
2. Uncontrolled infection;patients with positive HBsAg or HBcAb and peripheral blood HBV DNA titer detection ≥ 1 × 10^2 copy number / L; HCV antibody positive and peripheral blood HCV RNA positive; HIV antibody positive; CMV DNA positive; syphilis positive;
3. Any instability of systemic disease, including but not limited to unstable angina, cerebrovascular accident, or transient cerebral ischemic (within 6 months prior to screening), myocardial infarction (within 6 months prior to screening), congestive heart failure (New York heart association (NYHA) classification ≥ III), need drug therapy of severe arrhythmia, liver, kidney, or metabolic disease;
4. Any uncontrolled disease may affect entry
5. Current or history of CNS involvement by malignancy.Known history or presence of clinically relevant central nervous system (CNS) pathology. Patients with a known history or prior diagnosis other immunologic or inflammatory disease affecting the CNS (such as epilepsy)
6. Patients who are receiving systemic steroid treatment and requiring long-term systemic steroid treatment during the treatment as determined by the investigator before screening (except inhalation or topical use); And subjects treated with systemic steroids (except inhalation or topical use) within 72h prior to cell transfusion;
7. Pregnant or lactating woman, and female subject who plans to have a pregnancy within 1 year after cell transfusion, or male subject whose partner plans to have a pr egnancy within 1 year after cell transfusion;
8. Active or uncontrollable infection requiring systemic therapy
9. Received CAR-T treatment or other gene therapies before enrollment;
10. Kown be allergic to anti-TRBC1 CAR-T cells or drugs(Fludarabine or Cyclophophamide)
11. The investigators consider other conditions unsuitable for enrollment.
12. Patients who may not be able to sign the Informed Consent due to disease,or who do not understand or unwillingness or inability to comply with research requirements

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2021-03-31 (Actual); Primary Completion 2023-11-26 (Estimated); Study Completion 2023-11-26 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability | 28 days post infusion
  Safety measured by occurence of study related adverse effects defined by NCI CTCAE5.0

SECONDARY OUTCOMES:
CAR-T cell expansion and persistence | 2 years post infusion
  To evaluate anti-TRBC1 CAR-T cell expansion and persistence after infusion
Total response rate (ORR) after administration | 3 months post infusion
  CR+CRi for T-ALL CR+PR for T cell lyphoma
Duration of remission (DOR) after administration | 2 years post infusion
  Duration of remission (DOR) after administration
Overall Survival (OS)after administration | 2 years post infusion
  Overall Survival (OS)after administration
Progression Free Survival (PFS) after infusion | 2 years after infusion
  Progression Free Survival (PFS) after infusion

CONTACTS AND LOCATIONS:
Locations (1):
- Xianmin Song, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No